CLINICAL TRIAL: NCT02997046
Title: Use of Ferumoxytol Enhanced Magnetic Resonance Angiography for Cardiovascular Assessment in Late-stage Chronic Kidney Disease
Brief Title: Ferumoxytol Enhanced Magnetic Resonance Angiography in Chronic Kidney Disease
Acronym: FeMRA in CKD
Status: Completed | Type: Observational
Sponsor: Sokratis Stoumpos (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor-Investigator, Sokratis Stoumpos, Doctor, University of Glasgow
Organization: University of Glasgow (Other)
Other Study IDs: GN16RE117
Record Dates: First submitted 2016-12-14; First posted 2016-12-19 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Ferric Compounds; Magnetic Resonance Angiography; Vascular Grafting; Arteriovenous Fistula; Kidney Transplantation
Keywords: Ferumoxytol; MRI; fistula; graft; kidney transplant; angiography; arteriovenous
MeSH Terms: conditions — Arteriovenous Fistula; Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Pre-transplant assessment: * CTA abdominal and aortoiliac vasculature before transplantation
  * FeMRA abdominal and aortoiliac vasculature & CMR before transplantation
- Mapping & surveillance (for fistula): * US vascular mapping before fistula creation
  * 6 week US fistula arm
  * FeMRA fistula arm/central veins & CMR before fistula creation and at 6 weeks
- Mapping & surveillance (for graft): * US vascular mapping before graft creation
  * 6 week US graft arm
  * FeMRA fistula arm/central veins & CMR before graft creation and at 6 weeks

SUMMARY:
Conventional vascular imaging techniques are often either contra-indicated in chronic kidney disease (CKD) patients due to their relative invasiveness, risks and cost. Computed tomography angiography (CTA) requires radiation and nephrotoxic iodinated contrast which may precipitate significant worsening of renal function and even prompt the need for institution of dialysis. Magnetic resonance angiography (MRA) using gadolinium-based contrast agents has been associated with the rare disease nephrogenic systemic fibrosis. Alternative imaging methods also have drawbacks: for example, this frail patient group has a higher risk of complications from conventional invasive catheter-based angiography, non-contrast-enhanced MRA allows visualization of smaller arteries but is less accurate for larger vascular structures, and ultrasound is often not appropriate for evaluation of the deep vessels of the abdomen and pelvis.

Ferumoxytol is an ultrasmall superparamagnetic iron oxide particle encapsulated by a semisynthetic carbohydrate, which was initially developed as a magnetic resonance imaging (MRI) contrast agent in 2000. However, interest in ferumoxytol as a therapeutic agent for the treatment of iron deficiency anaemia in the setting of CKD eclipsed its use as MRI contrast agent. During the last decade, ferumoxytol has gained appeal as an MRI contrast agent in patients with estimated glomerular filtration rates <30mL/min and there are reports in the literature for its safe use and utility in both adult and pediatric patients with CKD.

Participants will be selected from those who have been referred for assessment prior to kidney transplant or prior to vascular access creation for haemodialysis and will be divided into three groups. The first group will include patients who will undergo a CTA of abdominal and aortoiliac vasculature as part of their preparation for potential kidney transplantation. The second and third groups will include patients who are having a fistula or a graft created for dialysis, respectively. These patients are routinely having US vascular mapping to visualise the blood vessels before a fistula or a graft is created. Additionally, patients included in the second and third groups are routinely having surveillance scans of their fistula or graft at 6 weeks following creation. Study participants undergoing standard imaging tests as part of their clinical care will also have ferumoxytol-enhanced MRA (FeMRA).

DETAILED DESCRIPTION:
This is a comparative study in a cohort of patients with significant renal impairment. Study participants undergoing standard imaging tests as part of their clinical care will also have FeMRA. The investigators will compare outcomes of interest including quality of image and diagnostic accuracy in a head-to-head design.

These hypotheses will be tested:

1. FeMRA is superior to CTA for characterisation of abdominal and aortoiliac anatomy (pre-transplant assessment) before implantation of a kidney graft as it can robustly evaluate both arterial and venous anatomy.
2. FeMRA is superior to Doppler US for characterisation of vascular anatomy (vascular mapping) before vascular access creation as it can robustly assess central vein patency.
3. FeMRA is superior to Doppler US for characterisation of fistula (or graft) arm vascular anatomy (surveillance) at 6 weeks after fistula creation.
4. Integrated cardiac and vascular assessment using FeMRA before vascular access creation can better predict outcomes.

Patients will be selected from those who have been referred for assessment prior to kidney transplant or prior to vascular access creation for haemodialysis and will be divided into 3 different groups. The first group (group A) will include patients who are having CTA of abdominal and aortoiliac vasculature performed for pre-transplant assessment. The other two groups will include patients who are having US vascular mapping performed before arteriovenous fistula (group B) or synthetic graft (group C) creation for haemodialysis. These patients are routinely having US Doppler of their fistula arm at 6 weeks following access creation for surveillance. FeMRA will be performed in addition to standard care, i.e. patients in group A will have a single FeMRA at baseline while patients in groups B and C will have a FeMRA at baseline and a second one at 6 weeks. All patients will undergo Cardiac MR with Ferumoxytol at the same time. This is to assess whether cardiac parameters before transplantation or access creation are associated with outcomes (baseline Cardiac MR). The 6-weeks Cardiac MR aims to assess cardiovascular functional parameters (blood flow, cardiac output, systolic and diastolic function) after vascular access creation.

Imaging will be performed on a 3T Prisma (Siemens) MRI system. A total dose of 3mg of Ferumoxytol/kg of patient weight will be delivered but not to exceed one vial (510mg). In all cases Ferumoxytol will be diluted to a concentration no greater than 1 part Ferumoxytol to 4 parts 0.9% sodium chloride and will be administered with several spaced infusions of diluted agent for the different imaging components. Ferumoxytol infusion is controlled by a sophisticated MRI compatible infusion pump for precise control over infusion rate. This procedure would take a minimum of 20 minutes before the full cumulative dose is administered for a usual size patient and even longer for the maximum expected dose of 510 mg in a very large patient. As such the investigators are anticipating that patients will be scheduled for up to 45 minutes of imaging.

Small fractions of the dose will be administered initially as an infusion for myocardial perfusion and first pass imaging with a dynamic contrast enhanced (DCE) technique. After the full dose is administered, steady state high-resolution imaging will be undertaken using an ultrafast spoiled gradient echo sequences. Cardiac MR consisting of cardiac output, end systolic volume, end diastolic volume, aortic distensibility and flow Cardiac MR will be performed. Images will be obtained for left ventricular and right ventricular mass and function plus flow quantification.

The MRA will be reviewed by vascular radiology consultants (with between 6 and 20 years' experience) and a standard clinical report issued on the findings. At the end of the study, all imaging (US Doppler, CTA and investigatory MRA) will be jointly reviewed by the radiologists and other investigators in the study team. An independent radiologist that is not directly involved in the study will also review images. All discrepancies will be resolved by mutual consensus between the radiologists.

The general analytical approach will be to estimate accuracy (95% CI), sensitivity (95% CI) and specificity (95% CI) of FeMRA and standard imaging techniques. In addition, Cohen's κ with 95% CI will be computed to quantify the agreement between the FeMRA and standard imaging findings. A value of κ>0.7 indicates a high level of agreement. Because multiple image locations from each patient will be used for the statistical evaluation (at least 20 vascular cross sections from each scan), the interdependence of each location for a given patient examination will be assessed by use of a κ statistic. A value of κ<0.4 indicates weak or no interdependence. The investigators aim to recruit 20 patients in group A and 10 patients in each of the other two groups. Assuming that FeMRA will identify 10% more clinically significant vascular anatomic characteristics compared with CTA/US, then one would need to study 180 vascular sections in total to show a significant difference between tests using chi-squared test, assuming power of 80% and probability of type 1 error of 5%.

To evaluate associations between anatomical predictor variables and outcomes, multiple linear and logistic mixed-effects regression models will be used. Associations of fistula and graft outcomes with predictors will be treated as uniform across all anatomical configurations unless there is strong statistical or biological evidence to suggest otherwise. Based on data from a retrospective study performed at the same centre, the investigators assume a fistula failure rate of 30%.

ELIGIBILITY:
Inclusion Criteria:

1. Planned surgical creation of an autogenous upper-extremity fistula or synthetic graft.

   AND Current treatment with maintenance haemodialysis or anticipated treatment with maintenance haemodialysis within 6 months after planned fistula or graft creation surgery.

   OR Planned imaging of abdominopelvic vasculature as part of pre-transplant assessment.
2. Anticipated ability to comply with study procedures.
3. Ability to provide informed consent.

Exclusion Criteria:

1. Life expectancy ≤6 months.
2. Frail, elderly patients with multiple or serious co-morbidities (doctor's discretion).
3. Pregnancy, lactation or women of child-bearing potential not willing to use effective contraception for the duration of the study.
4. Standard contra-indications to MRI and severe claustrophobia.
5. History of allergic reaction to any intravenous iron product, known hypersensitivity to excipients, asthma, eczema, atopy, patients with immune or inflammatory conditions (e.g. systemic lupus, rheumatoid arthritis), any conditions associated with iron overload (e.g. haemochromatosis, chronic liver disease, or blood disorders requiring frequent blood transfusions), and known history of drug allergy.
6. Any other reason considered by a study physician to make subject inappropriate for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Comparison of FeMRA with standard imaging techniques in assessment of vascular anatomy. | Baseline and week 6
  Multiple cross sections of various vascular beds obtained with currently used imaging techniques will be compared with matched sections obtained with FeMRA in a blinded fashion. The emphasis is generally on imaging quality and diagnostic accuracy on identification of clinically significant anatomic characteristics or lesions.

SECONDARY OUTCOMES:
Comparison of FeMRA with standard imaging techniques in identification of anatomical predictors of vascular access outcomes. | Up to 2 years
  Outcomes include:
  1. Sonographic anatomical fistula maturation at 6 weeks after creation.
     Criteria of sonographic AVF maturation include:
     * AVF lumen diameter >4mm and
     * AVF blood flow >500mL/min
  2. Fistula or graft complications: stenosis, thrombosis, hand ischaemia, aneurysm or pseudoaneurysm, infiltration, fistula bleeding, and infection.
  3. Fistula or graft procedures: surgical revision, angioplasty, stent placement, thrombolysis or thrombectomy, ligation of accessory veins, superficialisation of vein, transposition of vein, central venous catheter use, and placement of new arteriovenous access.
Association between cardiac function and fistula (or graft) outcomes assessed by FeMRA. | Up to 2 years
Effect of successful fistula (or graft) creation on cardiac function assessed by FeMRA. | Week 6
Utility of FeMRA in assessment of cardiac anatomy and function before listing for kidney transplantation. | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
No plans for sharing any data at the moment.

REFERENCES:
- [Derived] Stoumpos S, Tan A, Hall Barrientos P, Stevenson K, Thomson PC, Kasthuri R, Radjenovic A, Kingsmore DB, Roditi G, Mark PB. Ferumoxytol MR Angiography versus Duplex US for Vascular Mapping before Arteriovenous Fistula Surgery for Hemodialysis. Radiology. 2020 Oct;297(1):214-222. doi: 10.1148/radiol.2020200069. Epub 2020 Jul 21. PMID 32692301